CLINICAL TRIAL: NCT02312128
Title: Early Mobilization of Operatively Stabilized Distal Radius Fractures - a Randomized Controlled Trail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig Boltzmann Gesellschaft (Other)
Collaborators: Ludwig Boltzmann Institute for Traumatology - The research center in cooperation with AUVA (Other Government)
Responsible Party: Principal Investigator, Stefan Quadlbauer, M.D., M.D., AUVA Traumazentrum Vienna Site UKH Meidling
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03/2010
Record Dates: First submitted 2014-12-01; First posted 2014-12-09 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Closed Fracture of Lower End of Radius and Ulna
Keywords: distal radius fractures; early mobilization; postoperative treatment; outcome
MeSH Terms: conditions — Wrist Fractures | interventions — Surveys and Questionnaires; X-Rays; Hand Strength

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Mobilisation (Active Comparator): receives a removable plastic cast for one week and is allowed to move the wrist directly postoperative.
  Interventions:
  * Range of Motion measurement (ROM),
  * Grip strength measurement,
  * VAS Score according to the visual analogue scale ().
  * Questionnaire: PRWE Score, DASH Score and Mayo Wrist Score.
  * X- Rays in two planes.
  Follow-up: 6., 9., 12. postoperative week, a half and one year after surgery
  Interventions: Other: Questionnaire; Radiation: X- Ray; Other: Grip Strength; Other: VAS Score; Other: Range of Motion measurement
- Cast Group (Active Comparator): receives a non removable cast for 5 weeks
  Interventions:
  * Range of Motion measurement (ROM),
  * Grip strength measurement,
  * VAS Score according to the visual analogue scale ().
  * Questionnaire: PRWE Score, DASH Score and Mayo Wrist Score.
  * X- Rays in two planes.
  Follow-up: 6., 9., 12. postoperative week, a half and one year after surgery
  Interventions: Other: Questionnaire; Radiation: X- Ray; Other: Grip Strength; Other: VAS Score; Other: Range of Motion measurement

INTERVENTIONS:
Other: Questionnaire — DASH Score, PRWE Score, Mayo Wrist Score
Radiation: X- Ray — X-ray exposures in two planes 6., 9., 12. postoperative week, half and one year after surgery
Other: Grip Strength — Grip strength measurement
Other: VAS Score — Measurement pain according to the visual analogue scale (VAS)
Other: Range of Motion measurement — Angle measurement of the active range of motion in the wrist

SUMMARY:
The purpose of this study is to evaluate if an early mobilization after distal radius fractures treated by surgery leads to an better functional outcome then immobilization after surgery for 5 weeks in a cast

DETAILED DESCRIPTION:
All patients with a distal radius fracture treated by surgery (palmar angle stable plate) will be included in this study and randomised into two groups according the CONSORT Guidelines of Prospective Randomised Trails. One group ("early mobilisation") receive a removable plastic cast for one week and are allowed to move the wrist directly postoperative.

The other group ("control group") received a non removable cast for 5 weeks. Both groups underwent physiotherapy two times a week. The control group was only allowed to move the closed-by joints.

In the 6., 9., 12. postoperative week, a half and one year after the operation the patients underwent range of motion (ROM), grip strength measurement and pain according to the visual analogue scale (VAS). Hand function will be analysed according the PRWE (Patient-Rated Wrist Evaluation) Score, DASH (Disabilities of the Arm, Shoulder and Hand) Score and Mayo Wrist Score.

* Inclusion criteria:

  * Age ≥ 18 and ≤ 75 years
  * A2 - C3 distal radius fracture
  * no acute or older injury that influences hand function
  * operative stabilized by palmar angle stable plate
* Exclusion criteria:

  * Age ≥ 76 years
  * Age < 18 years
  * C3.3 radius fracture
  * acute or preexisting injures that influences hand function
  * pregnancy
  * neurologic disorders
  * incapacitated people

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years
* A2 - C3 distal radius fracture
* no acute or older injury that influences hand function
* operative stabilized by palmar angle stable plate

Exclusion Criteria:

* Age ≥ 76 years
* Age < 18 years
* C3.3 radius fracture
* acute or preexisting injures that influences hand function pregnancy neurologic disorders incapacitated people

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Functional Outcome as measured by visual analogue scale (VAS) | one year
  Pain evaluation according the VAS Score
Functional Outcome as measured by Range of Motion (ROM) | one year
  Range of Motion measured in sagittal plane, frontal plane and forearm rotation
Functional Outcome as measured by Patient - Rated Wrist Evaluation Score Patient - Functional Outcome as measured by Rated Wrist Evaluation (PRWE) Score | one year
  Questionnaire: PRWE Score
Functional Outcome as measured by Disabilities of the Arm, Shoulder and Hand (DASH) Score | One Year
  Questionnaire: DASH Score
Functional Outcome as measured by Mayo Wrist Score | One year
  Questionnaire: Mayo Wrist Score
Radiological outcome as measured by X-Ray | One Year
  Radiological outcome in x-ray of the Wrist in two planes
Functional Outcome as measured by Grip Strength | one year

SECONDARY OUTCOMES:
change Range of motion | 6., 9., 12. week postsurgery, a half and one year after surgery
Change Pain | 6., 9., 12. week postsurgery, a half and one year after surgery
Change Disabilities of the Arm, Shoulder and Hand (DASH) Score | 6., 9., 12. week postsurgery, a half and one year after surgery
Change Patient-Rated Wrist Evaluation (PRWE) Score | 6., 9., 12. week postsurgery, a half and one year after surgery
Change Mayo Wrist Score | 6., 9., 12. week postsurgery, a half and one year after surgery
Change X-Ray | 6., 9., 12. week postsurgery, a half and one year after surgery
  X-Ray of the wrist in two planes
Grip strength | 6., 9., 12. week postsurgery, a half and one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Quadlbauer, M.D., Principal Investigator — AUVA Traumazentrum Vienna Site UKH Meidling; Martin Leixnering, M.D., Study Director — AUVA Traumazentrum Vienna Site UKH Meidling
Locations (1):
- Austrian Workers' Compensation Board Trauma Hospital Lorenz Böhler, Vienna, Austria